CLINICAL TRIAL: NCT06522295
Title: Assessment of Optic Nerve Sheath Diameter in Preeclamptic Pregnant Women Using Ultrasonography and Anesthetic Management
Status: Not yet recruiting | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Tulay Sahin, professor, Kocaeli University
Other Study IDs: POSK23
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Preeclampsia; Intracranial Pressure Increase; Pregnancy; Anesthesia, Adverse Effect, Central Nervous System
MeSH Terms: conditions — Pre-Eclampsia; Intracranial Hypertension | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preeclampsia
  Interventions: Device: ultrasonography
- severe preeclampsia
  Interventions: Device: ultrasonography

INTERVENTIONS:
Device: ultrasonography — Ultrasonographic Measurement of Optic Nerve Sheath Diameter

SUMMARY:
Preeclampsia is a serious condition associated with complications such as pulmonary edema, placental abruption, hemolysis, thrombocytopenia, and cardiac, renal, and neurological complications, occurring at a rate of 2.7-8% in pregnant women (1,2). Neurological complications are believed to be associated with reversible cerebral vasoconstriction syndrome (3,4) and/or posterior leukoencephalopathy syndrome (4,5,6), sharing a common pathophysiology. Cerebral edema is primarily vasogenic, potentially linked to hyperperfusion resulting from impaired cerebral autoregulation, blood-brain barrier disruption, and endothelial cell dysfunction. In some eclampsia cases, computed tomography and magnetic resonance imaging may reveal signs consistent with significantly increased intracranial pressure (ICP) (7). However, the true incidence of elevated ICP in preeclampsia is unknown, clinical symptoms are nonspecific, and interpretation, especially during pregnancy and preeclampsia, can be challenging (2).

Cesarean section, currently one of the most frequently performed surgeries worldwide, is conducted in 21.1% of women (8). Anesthesia for cesarean section can be divided into neuraxial and general anesthesia. The choice of anesthesia technique in conditions that may increase intracranial pressure, such as cerebral edema, may vary based on balancing risks and benefits. Neuraxial analgesia and anesthesia are the first choice in healthy pregnancies, but may be contraindicated in cases with intracranial lesions or increased bleeding risk (9). The presence of focal neurological deficits may favor general anesthesia for cesarean delivery (10). General anesthesia in these patients may result in an increased hemodynamic response to laryngoscopy. Agents used in induction and maintenance can also affect cerebral autoregulation (11). Anesthesia induction and maintenance for these patients should be planned to minimize the increase in intracranial pressure.

The optic nerve, a part of the central nervous system, is surrounded by a dural sheath and a subarachnoid space containing cerebrospinal fluid. Three millimeters behind the ocular globe, the optic nerve is solely surrounded by fat, and the dural sheath can retract within its fatty environment, particularly in conditions of increased pressure in the cerebrospinal fluid (2). Recent clinical studies have reported that ultrasonographic measurements of the optic nerve sheath diameter (ONSD) are correlated with increased intracranial pressure symptoms and may serve as a non-invasive reliable indicator of ICP (12,13). Studies have reported high inter-observer reliability for ONSD measurements (14,15). ONSD measurement is easy, repeatable at the bedside, rapid, inexpensive, and does not involve radiation.

Compared to healthy pregnant women, preeclamptic women are considered to have higher intracranial pressure during the childbirth process. Anesthetic management for delivery in these women can be complex and controversial. The aim of this study is to evaluate ultrasonographic measurements of optic nerve sheath diameter during the perioperative period, independent of anesthesia management, in healthy and preeclamptic pregnant women undergoing cesarean section. We believe that these assessments will contribute to more reliable anesthesia planning for preeclamptic pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* asa 2-3 Individuals Aged 18 and Above Individuals with Gestational Age of 37 Weeks and Above pregnancy with health, mild preeclampsia, severe preeclampsia

Exclusion Criteria:

* Multiple pregnancies Fetal anomalies Patients with contraindications to ocular ultrasound (allergy to ultrasound gel, ocular injury or infection, facial fracture) Conditions known to increase cerebral pressure (idiopathic intracranial hypertension, brain tumor, recent history of brain trauma) Conditions potentially leading to edema (heart failure, glomerulonephritis or nephrotic syndrome, liver failure, malnutrition, hypothyroidism) Ophthalmic conditions that may affect optic nerve sheath diameter measurement (glaucoma, cataracts, previous eye surgery) Chronic hypertension

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant womens with preeclampsia
Study Population: pregnant womens with mild and severe preeclampsia
Sampling Method: Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2024-09-22 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The Difference in Optic Nerve Sheath Diameter Between Severe and Mild Preeclampsia | 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dubost C, Le Gouez A, Jouffroy V, Roger-Christoph S, Benhamou D, Mercier FJ, Geeraerts T. Optic nerve sheath diameter used as ultrasonographic assessment of the incidence of raised intracranial pressure in preeclampsia: a pilot study. Anesthesiology. 2012 May;116(5):1066-71. doi: 10.1097/ALN.0b013e318246ea1a. PMID 22258019
- [Background] Hinchey J, Chaves C, Appignani B, Breen J, Pao L, Wang A, Pessin MS, Lamy C, Mas JL, Caplan LR. A reversible posterior leukoencephalopathy syndrome. N Engl J Med. 1996 Feb 22;334(8):494-500. doi: 10.1056/NEJM199602223340803. PMID 8559202
- [Background] Anson JA, Vaida S, Giampetro DM, McQuillan PM. Anesthetic management of labor and delivery in patients with elevated intracranial pressure. Int J Obstet Anesth. 2015 May;24(2):147-60. doi: 10.1016/j.ijoa.2015.01.004. Epub 2015 Jan 19. PMID 25794413
- [Background] Finfer SR. Management of labour and delivery in patients with intracranial neoplasms. Br J Anaesth. 1991 Dec;67(6):784-7. doi: 10.1093/bja/67.6.784. PMID 1768551